CLINICAL TRIAL: NCT05460299
Title: Effects of Closed Kinetic Chain Exercises on Balance and Gait in People With Multiple Sclerosis: A Randomized Controlled Trial
Brief Title: Closed Kinetic Chain Exercises for Balance and Gait Rehabilitation for People With MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anas Radi Hassan Alashram (Other)
Responsible Party: Sponsor-Investigator, Anas Radi Hassan Alashram, Associate Professor, Middle East University
Organization: Middle East University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SREC/22/05/043
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telko plus conventional physical therapy (CPT) (Experimental): All patients received 15-minute CPT, three times a week, for four weeks. The patients in the experimental group received 15-minute Telko at the end of each CPT session.
  Interventions: Combination Product: Telko plus conventional physical therapy (CPT)
- Conventional physiotherapy (Active Comparator): All patients received 15-minute CPT, three times a week, for four weeks.
  Interventions: Combination Product: Telko plus conventional physical therapy (CPT)

INTERVENTIONS:
Combination Product: Telko plus conventional physical therapy (CPT) — All patients underwent about 15-minute CPT sessions 3 days a week for 4 weeks. The CPT intervention program consisted of closed kinetic chain exercises (squatting, hip bridge, lunge, and toe standing), 3 sets, 10 repetitions each and gait training (walking forward, backward, sidewalk, and between obstacles). Short breaks (1-5 minutes) were provided, depending on the patient tolerance. Before treatment, the skilled physical therapist was instructed about the duration, frequency, and content of therapy. The patients in the experimental group received additional lower extremities closed kinetic chain training using the Telko device. The participants train on Telko for 15 minutes using moderate resistance, 3 days a week for 4 weeks.
  Other Names: conventional physiotherapy

SUMMARY:
In total, 27 patients with MS (Expanded Disability Status Scale (EDSS) score equal to or less than 5.5) were randomly assigned to either Telko plus conventional physical therapy (CPT) experimental group (n=14) or the CPT control group (n=13). All patients received 15-minute CPT, three times a week, for four weeks. The patients in the experimental group received 15-minute Telko at the end of each CPT session. The outcome measures used were the Berg Balance Scale (BBS), 6-Minute Walk Test (6MWT), and Timed Up and Go (TUG) assessment.

DETAILED DESCRIPTION:
Participants were included in the present study with a confirmed diagnosis of MS, adults over 20 years of age, and the Expanded Disability Status Scale (EDSS) score equal to or less than 5.5. Exclusion criteria were having any neurologic or orthopaedic disorders that influenced the patients' motor function (e.g., stroke, fractures), severe cognitive impairments, and spasticity more than 4 based on MAS.

The patients were randomly allocated to either the lower extremities closed kinetic chain training (Telko) and conventional physiotherapy (CPT) experimental group or the CPT alone control group. Permuted block randomisation was used with a block size of 4, and treatment assignment was concealed using sealed envelopes. The randomisation sequence was generated using the statistical analysis software, MedCalc version.

Conventional physiotherapy (CPT) All patients underwent about 15-minute CPT sessions 3 days a week for 4 weeks. The CPT intervention program consisted of closed kinetic chain exercises (squatting, hip bridge, lunge, and toe standing), 3 sets, 10 repetitions each and gait training (walking forward, backward, sidewalk, and between obstacles). Short breaks (1-5 minutes) were provided, depending on the patient tolerance. Before treatment, the skilled physical therapist was instructed about the duration, frequency, and content of therapy.

Lower extremities closed kinetic chain training The patients in the experimental group received additional lower extremities closed kinetic chain training using the Telko device. The participants train on Telko for 15 minutes using moderate resistance, 3 days a week for 4 weeks.

Outcome measures The participants in both groups were clinically assessed at the baseline, the end of week 4 of treatment, and the 4-week follow-up by one assessor blinded to the intervention. Demographic information from each participant, including age, sex, body mass index (BMI), family history of MS, and the EDSS scores, was collected. The participants were assessed using the 6-minute walk test (6-MWT), Berg Balance Scale (BBS), and Timed-Up and Go (TUG).

The 6-MWT was used to assess functional capacity in people with MS (Goldman et al., 2008). It measures the distance covered by the patient in 6 minutes (Goldman et al., 2008). It is a good predictor of cardiorespiratory endurance in patients with MS (Goldman et al., 2008). The 6-MWT for people with MS has shown good reliability (ICC = 0.96-0.98) and good discriminant validity (Bartels et al., 2012; De Groot & Takken, 2011). The 6-MWT for people with MS has revealed good reliability (ICC = 0.96-0.98) and good validity (Bartels et al., 2012; De Groot & Takken, 2011). The test was administrated according to the guidelines provided by of American Thoracic Society (ATS) (ATS Statement, 2002). Two canes were placed 30 meters from each other. Before and immediately after the test, heart rate and oxygen saturation were documented using a pulse oximeter. The participant was able to complete the 6-MWT without taking a rest break. Gait speed was exhibited in meters per minute by dividing the total distance covered in the 6-MWT by 6 minutes.

Balance was evaluated using the BBS. It has excellent reliability (ICC = 0.986) in people with MS (Cattaneo et al., 2007). This scale contains 14 items instructing patients to complete tasks related to the everyday life of varying difficulty levels. A score of zero represents an inability to complete the task, and a score of 4 expresses the ability to complete the task independently. The total final scores range from 0 to 56. A total score of less than 45 implies balance impairment (Berg, 1989; Zwick et al., 2000).

The TUG is a simple test used to evaluate an individual's mobility and demands static and dynamic balance (Kear et al., 2017). It has excellent reliability (ICC = 0.98) in people with MS (Valet et al., 2019). It utilises the time that an individual takes to rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. During the test, the person is expected to wear their regular footwear and use any mobility aids that they would normally need. Scores of 10 seconds or less exhibit normal mobility, 11 - 20 seconds are within normal limits for disabled individuals, and greater than 20 seconds implies the individual needs aid outside and suggests additional examination and intervention (Kear et al., 2017). A score of 30 seconds or more points that the individual may be prone to falls (José Gonçalves et al., 2015).

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis
* Over 20 years of age
* Expanded Disability Status Scale (EDSS) score equal to or less than 5.5.

Exclusion Criteria:

* Neurologic or orthopaedic disorders (e.g., stroke, fractures)
* Severe cognitive impairments
* Spasticity more than 4 based on MAS.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-04 (Estimated); Primary Completion 2023-08-16 (Estimated); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test (6-MWT) | Change from baseline 6-minute walk test at 4-week
  The 6-MWT was used to assess functional capacity in people with MS (Goldman et al., 2008). It measures the distance covered by the patient in 6 minutes (Goldman et al., 2008). It is a good predictor of cardiorespiratory endurance in patients with MS (Goldman et al., 2008). The 6-MWT for people with MS has shown good reliability (ICC = 0.96-0.98) and good discriminant validity (Bartels et al., 2012; De Groot & Takken, 2011). The 6-MWT for people with MS has revealed good reliability (ICC = 0.96-0.98) and good validity (Bartels et al., 2012; De Groot & Takken, 2011). The test was administrated according to the guidelines provided by of American Thoracic Society (ATS) (ATS Statement, 2002). Two canes were placed 30 meters from each other. Before and immediately after the test, heart rate and oxygen saturation were documented using a pulse oximeter. The participant was able to complete the 6-MWT without taking a rest break.
Berg Balance Scale (BBS) | Change from baseline BBS at 4-week
  Balance was evaluated using the BBS. It has excellent reliability (ICC = 0.986) in people with MS (Cattaneo et al., 2007). This scale contains 14 items instructing patients to complete tasks related to everyday life of varying difficulty levels. A score of zero represents an inability to complete the task, and a score of 4 expresses the ability to complete the task independently. The total final scores range from 0 to 56. A total score of less than 45 implies balance impairment (Berg, 1989; Zwick et al., 2000).

SECONDARY OUTCOMES:
Timed-Up and Go (TUG) | Change from baseline TUG at 4-week
  The TUG is a simple test used to evaluate an individual's mobility and demands static and dynamic balance (Kear et al., 2017). It has excellent reliability (ICC = 0.98) in people with MS (Valet et al., 2019). It utilises the time that an individual takes to rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. During the test, the person is expected to wear their regular footwear and use any mobility aids that they would normally need. Scores of 10 seconds or less exhibit normal mobility, 11 - 20 seconds are within normal limits for disabled individuals, and greater than 20 seconds implies the individual needs aid outside and suggests additional examination and intervention (Kear et al., 2017). A score of 30 seconds or more points that the individual may be prone to falls (José Gonçalves et al., 2015).

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Padua, PhD, Study Director — Universita Telematica San Raffaele Roma Srl
Locations (1):
- Isra University, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No